CLINICAL TRIAL: NCT02503228
Title: Clinical Assessment of the Missouri Osteochondral Allograft Preservation System: Lifelong Registry
Brief Title: Clinical Registry Assessment of the Missouri Osteochondral Allograft Preservation System - MOPS
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, James Cook, William & Kathryn Allen Distinguished Chair in Orthopaedic Surgery, University of Missouri-Columbia
Other Study IDs: 2002628; 2003053 (Other: Registry IRB)
Record Dates: First submitted 2015-07-13; First posted 2015-07-20 (Estimated); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Symptomatic Osteochondral Defect(s); Cartilage, Meniscus, Ankle, Knee, Shoulder, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 100 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- MOPS: Transplanted tissue preserved using the MOPS method and obtained from one AATB-approved tissue bank
  Interventions: Procedure: Standard of care osteochondral and or meniscal allograft transplantation
- Standard Preservation: Transplanted tissue preserved using standard preservation methods and obtained from one of three AATB-approved tissue banks
  Interventions: Procedure: Standard of care osteochondral and or meniscal allograft transplantation

INTERVENTIONS:
Procedure: Standard of care osteochondral and or meniscal allograft transplantation — Standard of care osteochondral and or meniscal allograft transplantation

SUMMARY:
With institutional review board approval and informed consent, patients are prospectively enrolled into a registry to follow outcomes after osteochondral allograft (OCA) and/or meniscal allograft transplantation. Patients are included when 1 year followup data are available, including complications and reoperations, patient reported outcome measures (PROMs), compliance with rehabilitation, revisions, and failures.

In addition, MOPS grafts are compared to standard preservation grafts, and unipolar, multisurface, and bipolar cohorts, as well as patient compliance variables, are compared.

DETAILED DESCRIPTION:
With institutional review board approval and documented informed consent, patients are prospectively enrolled into a dedicated registry designed to follow outcomes after OCA transplantation with or without meniscal allograft transplantation. All grafts are obtained from tissue banks accredited by the American Association of Tissue Banks (AATB) and used in conformance of the tissue to the US Food and Drug Administration classification of a human cell and tissue product under section 361 of the Public Health Services Act. Initially, standard preservation (SP) grafts stored in refrigeration in proprietary solutions for 21 days after recovery from 1 of 3 AATB accredited tissue banks were used. As a separate arm, first clinical use of Missouri Osteochondral Preservation System (MOPS) grafts, which are stored at room temperature using MOPS methods for up to 56 days after recovery from 1 AATB accredited tissue bank, was assessed. In phase 2, after MOPS grafts became commercially available, type of graft implanted was based on patient-matched graft availability. Then, on the basis of emerging evidence published in the peer-reviewed medical literature, we implemented a shift in practice to discontinue use of SP grafts at our center.

Surgery is performed on patients with at least one large focal full-thickness articular cartilage defect and/or functional deficiency of 1 or both menisci for knee patients, and for hip, ankle or shoulder patients with at least 1 large focal full-thickness defect who chose this treatment option over other nonsurgical or surgical options as indicated and were approved for coverage by their insurance provider. OCA transplantation surgery is performed using press-fit cylindrical grafts and/or custom-cut patient-specific tab-in-slot shell grafts stabilized with either screws, bioabsorbable pins, or bioabsorbable nails. OCA bone is saturated with autogenous bone marrow aspirate concentrate (Angel System; Arthrex, Inc) immediately before implantation after subchondral drill holes are created and the donor bone is thoroughly lavaged to remove marrow elements. Meniscal allograft transplants (fresh or fresh frozen) are performed via a bone plug technique with suspensory fixation or included as part of the tibial OCA transplant. Viable chondrocyte density of OCAs at the time of transplantation are determined when tissues are available, as previously described. Procedure-specific postoperative management protocols are prescribed to each patient undergoing allograft transplantation. All patients receive oral and written instructions regarding postoperative rehabilitation.

Data are collected preoperatively and at 6 weeks, 3 months, 6 months, and yearly after surgery for each case. Demographic and operative data are collected from the electronic medical record. Patient-reported outcome measures (PROMs) are collected at each time point. All reported complications and reoperations are recorded in the electronic medical record. Revision is defined as a second operation to revise the osteochondral and/or meniscal allograft in at least 1 part of the patient's joint, and failure is defined as conversion to total or partial artificial joint arthroplasty, joint fusion, or amputation. The decision to pursue revision or failure surgery is based on the attending surgeon's discussion of joint pathology, treatment options, and related prognosis in conjunction with patient preference. Successful outcomes are defined as patients reporting return to functional activities with no need for revision or conversion surgery at last recorded follow-up. Descriptive statistics are calculated to report means, ranges, and percentages. On the basis of the difference in graft preservation methodology, cases are also analyzed by cohort as defined by SP versus MOPS. On the basis of surgery type, cases are also analyzed by cohort as defined by unipolar, multisurface, or bipolar transplants. Chi-square or Fisher exact tests are used to assess for significant differences in proportions. When significant differences in proportions are noted, odds ratios are calculated for relevant comparisons. One-way analysis of variance or t tests are used to assess for significant differences among cohorts at respective time points. Repeated measures analyses of variance are used to assess for significant differences within cohorts over time. Kaplan-Meier survival probability estimates with 95% CIs are calculated and compared. Significance is set at P<.05.

ELIGIBILITY:
Inclusion Criteria:

1. Adults and children age ≥13 years
2. Knee, hip, ankle, or shoulder osteochondral defect ≥15mm as determined by MRI or diagnostic knee arthroscopy for allograft transplantation
3. Must be physically and mentally willing and able to comply with postoperative and routinely scheduled clinical and radiographic evaluations.
4. Must be able to read and understand English or a language for which translated versions of the patient reported questionnaires and Informed consent form are available.
5. Must be able to sign informed consent and must voluntarily sign the Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved subject Informed Consent Form.

Exclusion Criteria:

1. Is a prisoner
2. Is receiving workman's compensation
3. Subject is mentally incompetent such that would preclude the subject from providing adequate consent and/or complying with study requirements

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients enrolled will be those that have undergone an OCA and or meniscal transplantation at University of Missouri Healthcare (Mizzou BioJoint Center) and consented to inclusion in the registry
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2050-12 (Estimated); Study Completion 2050-12 (Estimated)

PRIMARY OUTCOMES:
International Knee Documentation Committee (IKDC) | annually up to 29 years
  The International Knee Documentation Committee (IKDC) Subjective Knee Form is a patient-oriented questionnaire that assesses symptoms and function in daily living activities.
PROMIS survey (PROMIS Bank v1.2 - Physical Function) | annually up to 29 years
  PROMIS® stands for Patient Reported Outcomes Measurement Information System, which is a system of highly reliable, precise measures of patient-reported health status for physical, mental, and social well-being. In this particular case, this survey assesses the patient's physical function.
Visual Analogue Scale (VAS) Pain Score | annually up to 29 years
  The visual analog scale (VAS) is a tool widely used to measure pain. A patient is asked to indicate his/her perceived pain intensity (most commonly) along a 10 cm horizontal line, and this rating is then measured from the left edge (=VAS score)
Single Assessment Numeric Evaluation (SANE) | annually up to 29 years
  SANE is a patient rating from 0-100. Patients rate their current illness score in relation to their pre-injury baseline.
Success, Revision, Failure | annually up to 29 years
  Revision is defined as a second operation to revise the osteochondral and/or meniscal allograft in at least 1 part of the patient's joint, and failure is defined as conversion to artificial arthroplasty, arthrodesis, or amputation. Successful outcomes are defined as patients reporting return to functional activities with no revision or failure at last recorded follow-up.
PROMIS survey (PROMIS Bank v1.2 - Physical Function - Mobility | annually up to 29 years
  PROMIS® stands for Patient Reported Outcomes Measurement Information System, which is a system of highly reliable, precise measures of patient-reported health status for physical, mental, and social well-being. In this particular case, this survey assesses the patient's mobility.

SECONDARY OUTCOMES:
PROMIS survey (PROMIS Bank v1.1 - Pain Interference) | annually up to 29 years
  PROMIS® stands for Patient Reported Outcomes Measurement Information System, which is a system of highly reliable, precise measures of patient-reported health status for physical, mental, and social well-being. In this particular case, this survey assesses how the patient's pain interferes with their general life style.
Standard of Care (SOC) Diagnostic Imaging | Pre-operative, 6 week, 3 month, 6 month, and annually up to 29 years
  When the study patient attends their standard-of-care visits with their primary surgeon, the surgeon may or may not order diagnostic radiological imaging (X-Ray, MRI) depending on their medical judgment.
  If such radiological imaging is ordered and the images are available, they will be evaluated to assess the healing and integration of the graft.
Blood and Urine Samples | Pre-operative, Day of Surgery, 6 week, 3 month, 6 month, and annually up to 29 years
  Blood and urine samples will be collected pre-operatively, at each surgical procedure (at the initial surgical procedure and any necessary procedure thereafter), and at each post-operative visit after the initial 2 week visit (6 weeks, 3 months, 6 months, 12 months, 24 months). These samples will be used to evaluate biomarkers associated with tissue inflammation, synthesis, degradation, and cell death.
Non-SOC MRI | 12 month visit
  A non-standard-of-care MRI will be taken at the 12 month visit to assess the healing and integration of the graft.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri, Columbia, Missouri, United States

REFERENCES:
- [Background] Schreiner AJ, Stannard JP, Stoker AM, Bozynski CC, Kuroki K, Cook CR, Cook JL. Unicompartmental bipolar osteochondral and meniscal allograft transplantation is effective for treatment of medial compartment gonarthrosis in a canine model. J Orthop Res. 2021 May;39(5):1093-1102. doi: 10.1002/jor.24801. Epub 2020 Jul 27. PMID 32672863
- [Background] Thomas DM, Stannard JP, Pfeiffer FM, Cook JL. Biomechanical Properties of Bioabsorbable Fixation for Osteochondral Shell Allografts. J Knee Surg. 2020 Apr;33(4):365-371. doi: 10.1055/s-0039-1677837. Epub 2019 Feb 6. PMID 30727021
- [Background] Cook JL. Editorial Commentary: Bone Marrow Aspirate Biologics for Osteochondral Allografts-Because We Can or Because We Should? Arthroscopy. 2019 Aug;35(8):2445-2447. doi: 10.1016/j.arthro.2019.04.018. PMID 31395184
- [Background] Baumann CA, Baumann JR, Bozynski CC, Stoker AM, Stannard JP, Cook JL. Comparison of Techniques for Preimplantation Treatment of Osteochondral Allograft Bone. J Knee Surg. 2019 Jan;32(1):97-104. doi: 10.1055/s-0038-1636834. Epub 2018 Mar 7. PMID 29514363
- [Background] Cook JL, Stannard JP, Stoker AM, Bozynski CC, Kuroki K, Cook CR, Pfeiffer FM. Importance of Donor Chondrocyte Viability for Osteochondral Allografts. Am J Sports Med. 2016 May;44(5):1260-8. doi: 10.1177/0363546516629434. Epub 2016 Feb 26. PMID 26920431
- [Background] Cook JL, Stoker AM, Stannard JP, Kuroki K, Cook CR, Pfeiffer FM, Bozynski C, Hung CT. A novel system improves preservation of osteochondral allografts. Clin Orthop Relat Res. 2014 Nov;472(11):3404-14. doi: 10.1007/s11999-014-3773-9. Epub 2014 Jul 17. PMID 25030100
- [Background] Crist BD, Stoker AM, Pfeiffer FM, Kuroki K, Cook CR, Franklin SP, Stannard JP, Cook JL. Optimising femoral-head osteochondral allograft transplantation in a preclinical model. J Orthop Translat. 2015 Nov 25;5:48-56. doi: 10.1016/j.jot.2015.10.001. eCollection 2016 Apr. PMID 30035074
- [Background] Garrity JT, Stoker AM, Sims HJ, Cook JL. Improved osteochondral allograft preservation using serum-free media at body temperature. Am J Sports Med. 2012 Nov;40(11):2542-8. doi: 10.1177/0363546512458575. Epub 2012 Sep 12. PMID 22972852
- [Background] Stoker AM, Stannard JP, Kuroki K, Bozynski CC, Pfeiffer FM, Cook JL. Validation of the Missouri Osteochondral Allograft Preservation System for the Maintenance of Osteochondral Allograft Quality During Prolonged Storage. Am J Sports Med. 2018 Jan;46(1):58-65. doi: 10.1177/0363546517727516. Epub 2017 Sep 22. PMID 28937783
- [Background] Luk J, Stoker AM, Teixeiro E, Kuroki K, Schreiner AJ, Stannard JP, Wissman R, Cook JL. Systematic Review of Osteochondral Allograft Transplant Immunology: How We Can Further Optimize Outcomes. J Knee Surg. 2021 Jan;34(1):30-38. doi: 10.1055/s-0040-1721670. Epub 2021 Jan 3. PMID 33389738
- [Background] Nuelle CW, Nuelle JA, Cook JL, Stannard JP. Patient Factors, Donor Age, and Graft Storage Duration Affect Osteochondral Allograft Outcomes in Knees with or without Comorbidities. J Knee Surg. 2017 Feb;30(2):179-184. doi: 10.1055/s-0036-1584183. Epub 2016 May 26. PMID 27228198
- [Background] Stoker AM, Baumann CA, Stannard JP, Cook JL. Bone Marrow Aspirate Concentrate versus Platelet Rich Plasma to Enhance Osseous Integration Potential for Osteochondral Allografts. J Knee Surg. 2018 Apr;31(4):314-320. doi: 10.1055/s-0037-1603800. Epub 2017 Jun 24. PMID 28646824
- [Result] Stoker AM, Caldwell KM, Stannard JP, Cook JL. Metabolic responses of osteochondral allografts to re-warming. J Orthop Res. 2019 Jul;37(7):1530-1536. doi: 10.1002/jor.24290. Epub 2019 Mar 28. PMID 30912859
- [Result] Rucinski K, Cook JL, Crecelius CR, Stucky R, Stannard JP. Effects of Compliance With Procedure-Specific Postoperative Rehabilitation Protocols on Initial Outcomes After Osteochondral and Meniscal Allograft Transplantation in the Knee. Orthop J Sports Med. 2019 Nov 22;7(11):2325967119884291. doi: 10.1177/2325967119884291. eCollection 2019 Nov. PMID 31803790
- [Result] Zitsch BP, Stannard JP, Worley JR, Cook JL, Leary EV. Patient-Reported Outcomes for Large Bipolar Osteochondral Allograft Transplantation in Combination with Realignment Osteotomies for the Knee. J Knee Surg. 2021 Sep;34(11):1260-1266. doi: 10.1055/s-0040-1710361. Epub 2020 May 5. PMID 32369842
- [Result] Oladeji LO, Cook JL, Stannard JP, Crist BD. Large fresh osteochondral allografts for the hip: growing the evidence. Hip Int. 2018 May;28(3):284-290. doi: 10.5301/hipint.5000568. Epub 2017 Oct 17. PMID 29048690
- [Result] Stannard JP, Cook JL. Prospective Assessment of Outcomes After Primary Unipolar, Multisurface, and Bipolar Osteochondral Allograft Transplantations in the Knee: A Comparison of 2 Preservation Methods. Am J Sports Med. 2020 May;48(6):1356-1364. doi: 10.1177/0363546520907101. Epub 2020 Mar 5. PMID 32134685
- [Result] Rucinski K, Stannard JP, Crecelius C, Cook JL. Changes in knee range of motion after large osteochondral allograft transplantations. Knee. 2021 Jan;28:207-213. doi: 10.1016/j.knee.2020.12.004. Epub 2021 Jan 5. PMID 33418396
- [Result] Oladeji LO, Stannard JP, Cook CR, Kfuri M, Crist BD, Smith MJ, Cook JL. Effects of Autogenous Bone Marrow Aspirate Concentrate on Radiographic Integration of Femoral Condylar Osteochondral Allografts. Am J Sports Med. 2017 Oct;45(12):2797-2803. doi: 10.1177/0363546517715725. Epub 2017 Jul 24. PMID 28737949
- [Result] Stoker AM, Stannard JP, Cook JL. Chondrocyte Viability at Time of Transplantation for Osteochondral Allografts Preserved by the Missouri Osteochondral Preservation System versus Standard Tissue Bank Protocol. J Knee Surg. 2018 Sep;31(8):772-780. doi: 10.1055/s-0037-1608947. Epub 2017 Dec 11. PMID 29228404
- [Result] Cook JL, Rucinski K, Crecelius CR, Ma R, Stannard JP. Return to Sport After Large Single-Surface, Multisurface, or Bipolar Osteochondral Allograft Transplantation in the Knee Using Shell Grafts. Orthop J Sports Med. 2021 Jan 22;9(1):2325967120967928. doi: 10.1177/2325967120967928. eCollection 2021 Jan. PMID 33553437

DOCUMENTS (2):
  • Study Protocol (2015-07-14): https://cdn.clinicaltrials.gov/large-docs/28/NCT02503228/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-23): https://cdn.clinicaltrials.gov/large-docs/28/NCT02503228/SAP_001.pdf